CLINICAL TRIAL: NCT06686407
Title: Management of Lumbar Foraminal Stenosis Using Unilateral Biportal Endoscopy Versus Conventional Open Spine Surgery
Brief Title: Comparative Study Between Lumbar Foraminal Stenosis Treatment Modalities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Eldeen Mohamed Oreaby Adam, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lumbar Foraminal Stenosis
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Foraminal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Procedure: Open lumbar decompression ± fusion
- Group 2 (Experimental)
  Interventions: Procedure: Minimally invasive lumbar foraminal decompression using unilateral biportal endoscopy "device"

INTERVENTIONS:
Procedure: Open lumbar decompression ± fusion — Open lumbar decompression by laminectomy and transpedicular screw fixation using screws and rods ± interbody cage "device"
  Arms: Group 1
Procedure: Minimally invasive lumbar foraminal decompression using unilateral biportal endoscopy "device" — A new endoscopic technique that uses a Unilater Biportal Endoscopy for lumbar foraminal decompression
  Arms: Group 2

SUMMARY:
The goal of this clinical trial is to compare the clinical and radiological outcome of two different interventional techniques in lumbar foraminal stenosis decompression. The main questions it aims to answer are:

Does minimally invasive techniques give better results than conventional techniques?

Participants will:

Undergo minimally invasive intervention using unilateral biportal endoscopy for lumbar foraminal stenosis decompression Undergo lumbar fusion for lumbar foraminal stenosis decompression Keep a diary of their symptoms and improvement of these symptoms

DETAILED DESCRIPTION:
Lumbar foraminal stenosis decompression will be done using two different techniques:

1. Conventional Open Lumbar fusion By laminectomy and facetectomy and fixation with screws and rods ± interbody cage
2. Minimally invasive (Unilateral Biportal Endoscopy) Basic spine surgery instruments, 0° and 30° angled 4-mm diameter endoscopes commonly used in joint arthroscopic surgery, a radiofrequency catheter, Arthroscopic burr, and a shaver.

Surgical approach to the foraminal area Two portals are created to perform this surgery. Water is infused through the endoscope through the viewing portal, and the working portal had an additional purpose as a portal for water outflow. The proximal and distal portals are created 2 cm lateral from the pedicle level on the C-arm anteroposterior image. Each incision for the portals is 0.8 cm in length, which is adequate for instrument and endoscope insertion. For the left side foramen, the proximal and distal portals are used as the viewing and working portals, respectively, and vice versa for the right foramen. After the endoscope insertion through the viewing portal, we secure a space for the lower transverse process around the lateral surface of the facet joint. A radiofrequency catheter or a shaver is used to secure the space, and a radiofrequency catheter is used to control active bleeding.

Decompression of foraminal stenosis After a sufficient working space is obtained, the cranial 50% of the superior articular process of the thickened facet joint is removed using an arthroscopic burr or an osteotome. After removing the superior articular process, the ligamentum flavum around the foramen is removed using a curette and a Kerrison punch. After completion of flavectomy, nerve root and epidural fat are identified. If herniated disc material is found preoperatively, additional discectomy is performed usually from the axilla of the root. Surgery is confirmed to be completed after achieving an amount of free space concordant with the diameter of the nerve root in the foraminal zone, and then a drain tube is inserted.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with degenerative lumbar foraminal stenosis, diagnosed in outpatient clinic.
* Patients (age >18 )

Exclusion Criteria:

* Deformity.
* Infection of vertebrae.
* Tumor of vertebrae.
* Instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index (ODI) | Through study completion, an average of 2 years
Visual analogue scale (VAS) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Post operative radiological assessment by MRI on lumbosacral spine. | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wael Mohamed Ali, Assistant Professor, Study Director — Assiut University; Ahmed Hussein Mohamed, Lecturer, Study Director — Cairo University

REFERENCES:
- [Background] Kunogi J, Hasue M. Diagnosis and operative treatment of intraforaminal and extraforaminal nerve root compression. Spine (Phila Pa 1976). 1991 Nov;16(11):1312-20. doi: 10.1097/00007632-199111000-00012. PMID 1750006
- [Background] Lee S, Lee JW, Yeom JS, Kim KJ, Kim HJ, Chung SK, Kang HS. A practical MRI grading system for lumbar foraminal stenosis. AJR Am J Roentgenol. 2010 Apr;194(4):1095-8. doi: 10.2214/AJR.09.2772. PMID 20308517
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Soliman HM. Irrigation endoscopic decompressive laminotomy. A new endoscopic approach for spinal stenosis decompression. Spine J. 2015 Oct 1;15(10):2282-9. doi: 10.1016/j.spinee.2015.07.009. Epub 2015 Jul 10. PMID 26165475
- [Background] Hwa Eum J, Hwa Heo D, Son SK, Park CK. Percutaneous biportal endoscopic decompression for lumbar spinal stenosis: a technical note and preliminary clinical results. J Neurosurg Spine. 2016 Apr;24(4):602-7. doi: 10.3171/2015.7.SPINE15304. Epub 2016 Jan 1. PMID 26722954
- [Background] Choi DJ, Jung JT, Lee SJ, Kim YS, Jang HJ, Yoo B. Biportal Endoscopic Spinal Surgery for Recurrent Lumbar Disc Herniations. Clin Orthop Surg. 2016 Sep;8(3):325-9. doi: 10.4055/cios.2016.8.3.325. Epub 2016 Aug 10. PMID 27583117
- [Background] Storzer B, Schnake KJ. Microscopic bilateral decompression by unilateral approach in spinal stenosis. Eur Spine J. 2016 Aug;25 Suppl 2:270-1. doi: 10.1007/s00586-016-4479-3. No abstract available. PMID 26931328
- [Background] Poletti CE. Central lumbar stenosis caused by ligamentum flavum: unilateral laminotomy for bilateral ligamentectomy: preliminary report of two cases. Neurosurgery. 1995 Aug;37(2):343-7. doi: 10.1227/00006123-199508000-00025. PMID 7477792
- [Background] Bresnahan LE, Smith JS, Ogden AT, Quinn S, Cybulski GR, Simonian N, Natarajan RN, Fessler RD, Fessler RG. Assessment of Paraspinal Muscle Cross-sectional Area After Lumbar Decompression: Minimally Invasive Versus Open Approaches. Clin Spine Surg. 2017 Apr;30(3):E162-E168. doi: 10.1097/BSD.0000000000000038. PMID 28323694
- [Background] Guha D, Heary RF, Shamji MF. Iatrogenic spondylolisthesis following laminectomy for degenerative lumbar stenosis: systematic review and current concepts. Neurosurg Focus. 2015 Oct;39(4):E9. doi: 10.3171/2015.7.FOCUS15259. PMID 26424349
- [Background] Kim HJ, Jeong JH, Cho HG, Chang BS, Lee CK, Yeom JS. Comparative observational study of surgical outcomes of lumbar foraminal stenosis using minimally invasive microsurgical extraforaminal decompression alone versus posterior lumbar interbody fusion: a prospective cohort study. Eur Spine J. 2015 Feb;24(2):388-95. doi: 10.1007/s00586-014-3592-4. Epub 2014 Sep 25. PMID 25253301
- [Background] Hallett A, Huntley JS, Gibson JN. Foraminal stenosis and single-level degenerative disc disease: a randomized controlled trial comparing decompression with decompression and instrumented fusion. Spine (Phila Pa 1976). 2007 Jun 1;32(13):1375-80. doi: 10.1097/BRS.0b013e318064520f. PMID 17545903
- [Background] Chang SB, Lee SH, Ahn Y, Kim JM. Risk factor for unsatisfactory outcome after lumbar foraminal and far lateral microdecompression. Spine (Phila Pa 1976). 2006 May 1;31(10):1163-7. doi: 10.1097/01.brs.0000216431.69359.91. PMID 16648754
- [Background] Kovacs FM, Urrutia G, Alarcon JD. Surgery versus conservative treatment for symptomatic lumbar spinal stenosis: a systematic review of randomized controlled trials. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1335-51. doi: 10.1097/BRS.0b013e31820c97b1. PMID 21311394
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Ahmad S, Hamad A, Bhalla A, Turner S, Balain B, Jaffray D. The outcome of decompression alone for lumbar spinal stenosis with degenerative spondylolisthesis. Eur Spine J. 2017 Feb;26(2):414-419. doi: 10.1007/s00586-016-4637-7. Epub 2016 Jun 7. PMID 27272494
- [Background] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925
- [Background] Shenouda EF, Gill SS. Laminal fenestration for the treatment of lumbar nerve root foraminal stenosis. Br J Neurosurg. 2002 Oct;16(5):494-6; discussion 497. doi: 10.1080/0268869021000030320. PMID 12498495
- [Background] Ahn Y, Oh HK, Kim H, Lee SH, Lee HN. Percutaneous endoscopic lumbar foraminotomy: an advanced surgical technique and clinical outcomes. Neurosurgery. 2014 Aug;75(2):124-33; discussion 132-3. doi: 10.1227/NEU.0000000000000361. PMID 24691470
- [Background] Jenis LG, An HS. Spine update. Lumbar foraminal stenosis. Spine (Phila Pa 1976). 2000 Feb 1;25(3):389-94. doi: 10.1097/00007632-200002010-00022. PMID 10703115